CLINICAL TRIAL: NCT03674645
Title: Test and Optimization of New Specific MRI Sequences on an Imager Dedicated to Research
Acronym: SEQ-IRM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: L'Institut de RYthmologie et modélisation Cardiaque (IHU LIRYC) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2017/21
Record Dates: First submitted 2018-08-20; First posted 2018-09-17 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Magnetic Resonance Imaging Sequences
Keywords: Healthy volunteers; Test; Optimization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRI (Experimental): MRI exam performed on 200 healthy volunteers
  Interventions: Device: MRI acquisitions

INTERVENTIONS:
Device: MRI acquisitions — Procedure of the study is an MRI exam without any injection or invasive procedure, that will be performed on the Siemens Magnetom Aera imager of Liryc institute (L'Institut de RYthmologie et modélisation Cardiaque) (Xavier Arnozan site - Bordeaux)

SUMMARY:
Magnetic Resonance Imaging (MRI) performance depends on equipment performance, equipment maintenance and relevance of MRI sequence used. To optimize MRI performance, it's necessary to develop, optimize, test and validate new acquisition sequences for enhanced diagnosis and therapy monitoring. These new sequences will allow better spatial resolution and specificity while reducing acquisition time.

DETAILED DESCRIPTION:
The purpose of the present study is to test and optimize, on healthy subjects, specific MRI acquisition sequences firstly developed in a preclinical phase on phantoms (inert objects containing solutions or gels) and animal (Pig, sheep). This study will allow the investigators to define practical acquisition parameters that will allow reproducible results and precise definition of clinically relevant examination protocols for each new developed sequence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (over 18 yo),
* Male or female,
* Affiliated to social security,
* Without any contraindication to MRI exam and who will have signed a written inform consent.

Exclusion Criteria:

* Individuals deprived of liberty,
* Under guardianship or curatorship,
* Persons with known disease which could disturb MRI acquisition or with absolute or relative contraindication to an MRI examination
* Pregnant women,
* Breastfeeding women,
* Women without effective contraception,
* Participants who refused to be informed of the possible discovery of a significant anomaly,
* Persons involved in an interventional study with a drug or an implantable device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-09-19 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Image quality | Day 0
Signal to noise ratio | Day 0
Contrasts between structurally different regions | Day 0
  The values of the signal intensities will be measured in adjacent structures of interest. The difference between these values divided by the noise will be calculated to quantify the contrast-to-noise ratio between these structures. The higher this value is, the better is the sequence in its ability to differentiate these structures from one another.
Total acquisition time | Day 0
Qualitative interpretation of image quality to respiratory and cardiac motions | Day 0
  In the presence of improper compensation for cardiac and / or respiratory movements, the images may appear blurred. The qualitative interpretation of image quality will be performed by visual image analysis.
Quantitative interpretation of image quality to respiratory and cardiac motions | Day 0
  In the presence of improper compensation for cardiac and / or respiratory movements, the images may appear blurred. The quantitative interpretation of image quality will be performed by a measurement of sharpness of contours between adjacent structures of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Hubert COCHET, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Pessac, France

IPD SHARING:
Plan to Share IPD: No